CLINICAL TRIAL: NCT04593862
Title: Feasibility and Preliminary Efficacy of High-Intensity Interval Training in Bladder Cancer Patients Receiving Intravesical Therapy: a Randomized Controlled Trial
Brief Title: Bladder Cancer and ExeRcise Training During IntraVesical ThErapy
Acronym: BRAVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Northern Alberta Urology Centre (Unknown); Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HEBRA - CC 20-0184
Record Dates: First submitted 2020-10-02; First posted 2020-10-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Bladder Cancer
Keywords: Non-muscle invasive bladder cancer; Exercise; High-intensity interval training; Randomized Controlled Trial
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants and investigators will not be blinded to group assignment given the nature of the intervention. Outcome assessors will be blinded to group assignment for the clinical outcomes of tumour recurrence and progression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Group (Experimental): The exercise intervention will consist of 36 high-volume high-intensity interval sessions over a 12-week period. The exercise frequency will be three times per week during the 6 weeks of intravesical therapy and the 6 weeks of recovery (total 12 weeks) prior to a surveillance cystoscopy.
  Interventions: Other: High-Intensity Interval Training
- Usual Care: (No Intervention): Patients randomized to the control group will be asked not to initiate any exercise program or to increase their exercise level from baseline during the 12-week study. After the post-intervention assessments and 3-month cystoscopy, patients in the control group will be offered a 4-week supervised exercise program at the Behavioural Medicine Fitness Centre, University of Alberta.

INTERVENTIONS:
Other: High-Intensity Interval Training — The intervention will be performed on a treadmill and will include a warm-up and cool-down at 50-60% and 40% of the VO2peak respectively, for up to five minutes. The HIIT protocol will be 4x4, which consists of four bouts of four minutes at a workload corresponding to vigorous intensity (75-95% of the baseline and 6-week VO2peak) alternating with three minutes of recovery intervals at 40% of the VO2peak. The exercise session will last 35 minutes and include 16 minutes of high intensity exercise.
  Arms: Exercise Group

SUMMARY:
Bladder cancer is the fifth most common cancer in Canada and has the eighth highest cancer mortality rate. The treatment for the most frequent type of bladder cancer is surgically removing the tumour followed by six weeks of medication placed within the bladder. There are physical and psychosocial challenges from bladder cancer and its treatment that may affect how patients feel and function, and consequently their quality of life. Moreover, bladder cancer patients are at a high risk of their bladder cancer coming back and getting worse. Exercise is a low-cost intervention that may lower the chances of bladder cancer coming back or getting worse, manage side effects related to treatment, help patients feel better, and improve quality of life. To date, however, no study has examined if it is safe or even possible for bladder cancer patients to exercise when they are receiving drugs placed into their bladder. The Bladder cancer and exeRcise trAining during intraVesical thErapy (BRAVE) Trial will be the first study to test the safety, feasibility, and efficacy of exercise in bladder cancer patients during this drug therapy. The investigators will ask some patients to do a supervised exercise program during their drug treatment while other patients will be asked not to exercise. The investigators will compare the 2 groups on how they fare with their bladder cancer treatment. This study will provide information on whether exercise may help patients feel better, function better, and possibly even lower their chances of the disease coming back or getting worse.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will include men and women that (1) are ≥ 18 years old, (2) have a confirmed diagnosis of non-muscle invasive bladder cancer (clinical stage cis, Ta or T1), and (3) are scheduled to receive induction intravesical therapy with chemotherapy (e.g., Gemcitabine or Mitomycin) or immunotherapy (e.g., BCG) agents.

Exclusion Criteria:

* Exclusion criteria for participants include: (1) not being medically cleared to participate in the exercise intervention by their treating urologist and a certified exercise physiologist using the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+), (2) having contraindications for cardiopulmonary stress and/or physical fitness tests, (3) already exercising according to the Godin Leisure-Time Exercise Questionnaire (GLTEQ), (4) not having the ability to read and comprehend English, and (5) not willing to be randomized to a supervised exercise training program or usual care (no exercise) for 12 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Changes of Peak Oxygen Consumption (VO2peak) | At baseline, after the intravesical therapy (6-week), and 3-month follow-up
  VO2 peak will be directly measured by the modified Bruce treadmill protocol exercise test, using a metabolic measurement system system (Parvo Medics TrueOne® 2400; Sandy, UT, USA).VO2peak will be defined as the highest oxygen-uptake value recorded during the test and will be expressed as relative to body mass (i.e., ml O2·kg-1·min-1).

SECONDARY OUTCOMES:
Lower body strength | At baseline, after the intravesical therapy (6-week), and 3-month follow-up
  30-second chair stand
  Scores are compared with normative data based on sex and age, with "normal" defined as the middle 50% of the population. Those scoring above this range would be considered above average for their age and those below the range as below average
Upper body strength | At baseline, after the intravesical therapy (6-week), and 3-month follow-up
  Arm curl
  Scores are compared with normative data based on sex and age, with "normal" defined as the middle 50% of the population. Those scoring above this range would be considered above average for their age and those below the range as below average
Lower body Flexibility | At baseline, after the intravesical therapy (6-week), and 3-month follow-up
  Chair sit-and-reach
  Scores are compared with normative data based on sex and age, with "normal" defined as the middle 50% of the population. Those scoring above this range would be considered above average for their age and those below the range as below average
Upper body Flexibility | At baseline, after the intravesical therapy (6-week), and 3-month follow-up
  Back Scratch
  Scores are compared with normative data based on sex and age, with "normal" defined as the middle 50% of the population. Those scoring above this range would be considered above average for their age and those below the range as below average
Agility | At baseline, after the intravesical therapy (6-week), and 3-month follow-up
  8-foot up-and-go
  Scores are compared with normative data based on sex and age, with "normal" defined as the middle 50% of the population. Those scoring above this range would be considered above average for their age and those below the range as below average
Functional Capacity | At baseline, after the intravesical therapy (6-week), and 3-month follow-up
  6-minute walk test
  Scores are compared with normative data based on sex and age, with "normal" defined as the middle 50% of the population. Those scoring above this range would be considered above average for their age and those below the range as below average
Anthropometry and body composition measurements | At baseline, after the intravesical therapy (6-week), and 3-month follow-up
  Height, weight, waist, hip, and calf circumference
Health-related quality of life (HRQoL) | At baseline, 3-month (post-exercise intervention/prior to the 3-month surveillance cystoscopy), and at one-year follow-up
  Assessment of health-related quality of life (HRQoL) using the European Organization for Research and Treatment of Cancer (EORTC) core 30-item questionnaire (QLQ-C30) version 3.0.
  The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / quality of life scale, and six single items.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Bladder Cancer-Specific Quality of Life | At baseline, 3-month (post-exercise intervention/prior to the 3-month surveillance cystoscopy), and at one-year follow-up
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for non-muscle invasive bladder cancer core 24-item (EORTC QLQ NMIBC C24).
  EORTC QLQ NMIBC C24 is composed of scales assessing urinary symptoms, bowel symptoms, sexual, and side effects of intravesical treatment (fever, malaise, convenience of and worry due to repeated cystoscopies).
  All of the scales a range in score from 0 to 100. A high scale score represents a higher response level.
Fear of cancer recurrence/progression | At baseline, 3-month (post-exercise intervention/prior to the 3-month surveillance cystoscopy), and at one-year follow-up
  Fear of cancer recurrence/progression will be assessed by the Fear of Cancer Recurrence Inventory
  Minimum: 0 Maximum:168 Higher score= higher levels of fear of cancer recurrence/progression
Anxiety | At baseline, 3-month (post-exercise intervention/prior to the 3-month surveillance cystoscopy), and at one-year follow-up
  Anxiety will be assessed using the 10-item State-trait Anxiety Inventory.
  Minimum: 20 Maximum: 80 Higher score= worse anxiety
Depression | At baseline, 3-month (post-exercise intervention/prior to the 3-month surveillance cystoscopy), and at one-year follow-up
  Depression will be assessed using the Epidemiologic Studies Depression Scale (CES-D) questionnaire.
  Minimum: 0 Maximum: 30 (cut off point: 10) Higher score= worse depression
Perceived Stress | At baseline, 3-month (post-exercise intervention/prior to the 3-month surveillance cystoscopy), and at one-year follow-up
  Perceived stress will be assessed using the Perceived Stress Scale (PSS) questionnaire.
  questionnaire.
  Minimum: 0 Maximum: 56 Higher score=worse perceived stress
Fatigue | At baseline, 3-month (post-exercise intervention/prior to the 3-month surveillance cystoscopy), and at one-year follow-up
  Fatigue will be assessed using the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) questionnaire
  Minimum: 0 Maximum: 52 Higher score=worse fatigue
Self-esteem | At baseline, 3-month (post-exercise intervention/prior to the 3-month surveillance cystoscopy), and at one-year follow-up
  Self-esteem using the Rosenberg self-esteem scale
  Minimum: 10 Maximum: 40 Higher score= better self-esteem
Sleep quality | At baseline, 3-month (post-exercise intervention/prior to the 3-month surveillance cystoscopy), and at one-year follow-up
  Sleep quality will be assessed by the Insomnia Severity Index (ISI)
  Minimum: 0 Maximum: 28 Higher score= worse insomnia
Social cognitive predictors of exercise adherence: motivation, perceived benefits, enjoyment, support from others, self-efficacy, and barriers | At baseline, 3-month (post-exercise intervention/prior to the 3-month surveillance cystoscopy), and at one-year follow-up
  Standard scales for the Theory of Planned Behaviour

OTHER OUTCOMES:
Complete response | 3-month (post-exercise intervention/prior to the 3-month surveillance cystoscopy) and one-year follow-up
  Negative cytology, imaging, and cystoscopy and, when the TURBT is indicated, a negative biopsy.
Intravesical therapy adherence | 6-week follow-up
  Intravesical therapy adherence will be tracked by medical records of attendance and self-report drug retention time
Treatment toxicities | 6-week follow-up
  Treatment toxicities will be abstracted from medical records
Incidence of Adverse events related to the High-Intensity Interval Training during Intravesical Therapy | Through study completion, an average of 1 year
  To evaluate the safety of the program, any adverse events during the physical assessments (baseline, post- intravesical therapy, and post-intervention) and during the exercise sessions will be recorded.
Eligibility rate of non-muscle invasive bladder cancer patients to a high-intensity interval | At baseline
  The eligibility rate will be the number of non-muscle invasive bladder cancer patients
Recruitment rate of non-muscle invasive bladder cancer patients to a high-intensity interval training during Intravesical Therapy | At baseline
  The recruitment rate will be the number of non-muscle invasive bladder cancer patients enrolled in the study divided by the number of eligible patients.
Adherence rate of non-muscle invasive bladder cancer patients to a high-intensity interval | Through exercise intervention completion, an average of 12-weeks
  Adherence to the program will be measured by the number of exercise sessions completed without dose modifications. Reasons for not completing the exercise session or for dose adjustments will be recorded.
Follow-up assessment rate of non-muscle invasive bladder cancer patients to a high-intensity interval program during Intravesical Therapy | After the intravesical therapy (6-week), at the 3-month follow-up, and at 1 year follow-up
  The follow-up assessment rate will be determined by the number of participants who do not complete the post-intervention or follow-up assessments for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Kerry S Courneya, Principal Investigator — University of Alberta
Locations (1):
- Fernanda Zane Arthuso, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arthuso FZ, Fairey AS, Boule NG, Courneya KS. Bladder cancer and exeRcise trAining during intraVesical thErapy-the BRAVE trial: a study protocol for a prospective, single-centre, phase II randomised controlled trial. BMJ Open. 2021 Sep 24;11(9):e055782. doi: 10.1136/bmjopen-2021-055782. PMID 34561265